CLINICAL TRIAL: NCT07318012
Title: Impact of Isometric Handgrip Exercise Versus Walking on Blood Pressure: A Comparative Research Approach
Brief Title: Handgrip Exercise Versus Walking on Blood Pressure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Abubakr Mohamed Salama, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: handgrip exercise
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hypertensive Patients

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Isometric Handgrip Exercise
  Interventions: Procedure: Isometric Handgrip Exercise
- 2 (Experimental): Walking Exercise
  Interventions: Procedure: Walking Exercise
- 3 (No Intervention): Control Group

INTERVENTIONS:
Procedure: Isometric Handgrip Exercise — perform Isometric bilateral Handgrip Exercise
  Arms: 1
Procedure: Walking Exercise — Walking Exercise
  Arms: 2

SUMMARY:
The goal of this clinical study is to compare the effectiveness of isometric handgrip exercise versus walking exercise in improving blood pressure among hypertensive patients. The main question is Which of two exercise (Isometric Handgrip Exercise versus Walking Exercise) will be more effective in improvement Blood Pressure

ELIGIBILITY:
Inclusion Criteria:

stage 1 hypertension Medically stable

* Able to understand and follow instructions
* Willing to provide informed consent

Exclusion Criteria:

* • Stage 2 hypertension

  * Recent cardiovascular events
  * Uncontrolled diabetes mellitus
  * Severe orthopedic limitations
  * Neurological disorders
  * Pregnancy
  * Recent changes in antihypertensive medication (within 3 months)
  * Severe cardiac arrhythmias

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure measurment | 5 days
  decrease blood pressure measurement (systolic and dyastolic assessment)